CLINICAL TRIAL: NCT02138539
Title: A Clinical Usage Study to Evaluate the Safety and Efficacy of an Herbal-Based De-Pigmenting System
Brief Title: Evaluation of an Herbal-Based De-Pigmenting System
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sadick Research Group (Other)
Collaborators: Episciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SRG-EPI-1
Record Dates: First submitted 2014-02-26; First posted 2014-05-14 (Estimated); Last update posted 2015-11-18 (Estimated); Status verified 2015-11

CONDITIONS: Melasma; Hyperpigmentation
Keywords: hyperpigmentation; melasma; sun spots; dark spots
MeSH Terms: conditions — Melanosis; Hyperpigmentation | interventions — hydroquinone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 4% Hydroquinone (Active Comparator): 4% hydroquinone applied to one side of the face.
  Interventions: Drug: Hydroquinone
- Herbal depigmenting agent (Experimental): Herbal depigmenting agent applied on the other side of the face.
  Interventions: Other: Herbal depigmenting agent (Epionce)

INTERVENTIONS:
Other: Herbal depigmenting agent (Epionce) — A two product herbal pigmentation reducing regimen is applied twice a day to either the left or right side of the face for a duration of 4 months.
  Other Names: Epionce
  Arms: Herbal depigmenting agent
Drug: Hydroquinone — Hydroquinone 4% is applied twice a day to either the left or right side of the face for a duration of 4 months.
  Arms: 4% Hydroquinone

SUMMARY:
The purpose of this study is to evaluate the effectiveness and tolerability of an herbal de-pigmenting regimen applied to one side of the face compared with hydroquinone applied to the other side of the face in treating mottled hyperpigmentation and melasma.

DETAILED DESCRIPTION:
This clinical study is being conducted in order to evaluate the effectiveness and tolerability of a de-pigmenting regimen when used by subjects with mild to severe mottled hyperpigmentation and melasma. Efficacy will be assessed using visual grading, device measurements and digital photography. Tolerance and safety will be evaluated by grading for objective and subjective signs of irritation, and the incidence and severity of adverse events. Efficacy and tolerance of this product are compared to that of Hydroquinone, which is applied to one side of the subject's face while the herbal de-pigmenting regimen is applied to the other side of the face.

The two product pigmentation reducing herbal regimen is based on the novel concept of inhibiting all 14 major and the 3 branch steps in the melanin cascade.

ELIGIBILITY:
Inclusion Criteria:

* Female age 30-65
* Must be in good general health
* Must be willing to use sunscreen on the face daily
* Must be willing to avoid tanning beds and excessive exposure to direct sunlight
* Must be willing to continue using regular cosmetic regimen

Exclusion Criteria:

* Nursing pregnant/ planning to become pregnant during the course of the study
* Using a medication that increases sensitivity to sunlight including doxycycline, minocycline, tetracycline, ciprofloxin, hydrochlorothiazide, and sulfonamides.
* Any known allergies/sensitivities to facial skincare products, anti-aging products, de-pigmenting products, or products containing hydroquinone
* Usage of any new skincare products during the course of the study
* Presence of atopic dermatitis or psoriasis on the face
* Uncontrolled diabetes, hypertension, hypothyroidism, hyperthyroidism
* TCA or other deep peels within 1 year or medium to light peels within 3 months prior to starting the study
* Facial/laser treatment within the last 3 months
* Facial cosmetic surgery within the last 12 months
* Use of product, topical, or systemic medication, known to affect dyschromia, having "whitening" or anti-aging properties
* Physical skin conditions such as excessive hair, scarring, tattoos that might impair evaluations of the test sites
* Active hepatitis, immune deficiency, or autoimmune disease

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Melanin Index | 6 months
  The melanin index of the skin will be measured at baseline and at each follow-up visit with a non-invasive device. At the end of the study, the change of the Melanin index over a period of 6 months will be calculated.

SECONDARY OUTCOMES:
Irritation | Baseline, 1 month, 2 month, 4 month, 6 months
  Both objective irritation (erythema, edema, peeling, scaling/dryness) and subjective irritation (burning/stinging, itching, dry/tight feeling) will be measured at each visit via visual grading assessments and subject questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Neil S Sadick, MD, Principal Investigator — Sadick Research Group
Locations (1):
- Sadick Research Group, New York, New York, United States